CLINICAL TRIAL: NCT05320263
Title: Contact Aspiration Versus Stent Retriever for Recanalisation of Acute Stroke Patients With Basilar Artery Occlusion: The Posterior Circulation ASTER Randomized Trial
Brief Title: Contact Aspiration Versus Stent Retriever for Recanalisation of Acute Stroke Patients With Basilar Artery Occlusion: The Posterior Circulation ASTER Randomized Trial Protocol
Acronym: pc-ASTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_0105
Record Dates: First submitted 2022-02-14; First posted 2022-04-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Basilar Artery Occlusion
Keywords: Stroke; Basilar artery occlusion
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: It is planned to include a total of 480 patients (240 per am) to show with a 80% power an 12% increase in FPE rate at end of MT with contact aspiration technique, assuming 23 % of FPE in control arm, 5% of spontaneous recanalization and considering one interim futility analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contact aspiration first line thrombectomy (Experimental): Patient randomized in this arm will have the first arm thrombectomy by contact aspiration
  Interventions: Procedure: Contact aspiration Thrombectomy
- Stent retriever first line thrombectomy (Sham Comparator): Patient randomized in this arm will have the first arm thrombectomy by Stent retriever
  Interventions: Procedure: Stent retriever thrombectomy

INTERVENTIONS:
Procedure: Contact aspiration Thrombectomy — The contact aspiration approach is performed, as in standard care, using a long sheath positioned in the distal cervical vasculature using an exchange technique.
  A large bore balloon guide catheter as to be placed into the cervical ICA. The microcatheter is then advanced close to the thrombus and the large-bore aspiration catheter is advanced as close to the proximal aspect of the thrombus as possible. A control superselective angiogram may be used to document the extent of occlusion and thrombus. After a 3 min waiting period, the large-bore aspiration catheter is connected to a continuous aspiration from the dedicated aspiration pump while simultaneously advancing the aspiration catheter up to the face of the thrombus. through the long sheath positioned in the cervical vasculature.
  Arms: contact aspiration first line thrombectomy
Procedure: Stent retriever thrombectomy — The technique used should be in accordance with the device IFU. A large bore access guide catheter possible is recommended. A suitable delivery microcatheter is navigated over a microwire across the occlusion. A control superselective angiogram may be used to document the extent of occlusion and thrombus. The stent is left in place according to the internal practice of each participating center before the withdrawal. Any CE-marked stent retriever device is then deployed across the occlusion. A minimum of 3 attempts with SR should be performed. A revascularization score will be recorded after each device attempt.
  Arms: Stent retriever first line thrombectomy

SUMMARY:
Acute ischemic stroke (AIS) patients with basilar artery occlusion (BAO) present a devastating, life-threatening prognosis.

Urgent recanalization with endovascular mechanical thrombectomy is routinely performed in patients with BAO although the level of evidence is lower than that in anterior circulation occlusions (randomization in this population versus medical treatment alone having been impossible in recent studies). Recently, a large retrospective study supports the interest of thrombectomy in this population .

Speed and grade of the recanalisation have a major impact on clinical outcome. Favorable outcome at 90 days is strongly associated with the successful recanalization status at the end of the endovascular procedure (OR=4.57, 95%CI=1.24-16.87, P=0.023).

First pass effect has been shown to be a strong marker of efficacy of endovascular procedure with significant correlation with clinical outcome.

Thrombectomy with Stent retrievers dramatically changed the prognosis of anterior circulation large vessel occlusion strokes and currently used in BAO patients (posterior circulation). Contact aspiration (CA) is currently used in anterior large vessel occlusions (COMPASS trial, Lancet 2019), with similar rates of recanalization and favorable outcomes (Boulanger M, 2019), as well as in BAO patients .

However, the benefit of CA compared to SR for the treatment of BAO remains under debate with the superiority of first line CA compared to SR or no difference. Available data are based on retrospective studies with no data from RCT.

In this context, a randomized controlled trial is needed to assess the benefit of CA versus SR.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* AIS with BAO on non-invasive imaging (CT or MRI)
* Eligible for thrombectomy : groin puncture undergone within 24 hours of first symptoms or of last time the patient was seen normal
* Being covered by a national health insurance
* Informed consent obtained from the patients/his proxy or following an emergency procedure

Exclusion Criteria:

* Known or suspected pre-existing (chronic) large vessel stenosis / occlusion in the symptomatic territory (basilar artery)
* Severe contrast medium allergy or absolute contraindication to use of iodinated products
* Clinical history, past imaging or clinical judgment suggesting intracranial stenosis of the basilar artery
* Pregnancy (urine or serum beta HCG test for women of child-bearing potential)
* Person deprived of liberty
* Patient benefiting from a legal protection (guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-11-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of first pass effect (FPE) defined by complete reperfusion after first device pass | 24 hours
  The definition of FPE: single pass/use of the device, (2) complete revascularization of the large vessel occlusion and its downstream territory (mTICI 3), and (3) no use of rescue therapy

SECONDARY OUTCOMES:
Rate of complete reperfusion after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  mTICI (modified Thrombolysis In Cerebral Infarction ) score equals to 3 after the first line thrombectomy and at the end of endovascular.
  mTICI score is evaluated between 0-3 : 0 a complete obstruction of the artery and 3 indicates a complete reperfusion
Rate of successful reperfusion (mTICI 2b/2c/3) after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  mTICI score is evaluated between 0 to 3. Rate of patients with mTICI score equals to 2b/2c/3 after first-line thrombectomy strategy and at the end of endovascular procedure will be evaluated.
Rate of near to complete reperfusion (mTICI 2c/3) after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
Rate of Arterial Occlusive Lesion (AOL) recanalization score III after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  AOL recanalization score is evaluated between 0 to 3 :
  * 0 indicates no recanalization of the primary occlusive lesion
  * 3 indicates complete recanalization of the primary occlusive lesion with any distal flow
Groin puncture time to successful reperfusion time (evaluated in minutes) | 360 minutes
Modified Rankin Score (mRS) at 3 and 12 months | 12 months
  mRS is evaluated between 0 to 6. A score of 0 indicates that there is no disability and a score of 6 indicates death.
Rate of good functional outcome at 90-day and at one year defined by a mRS 0-3 or equal to pre-stroke mRS (Modified Rankin Score) | 12 months
Quality of life at 90 days and 12 months assessed by EuroQol 5D-5L scale | 12 months
  EuroQol 5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
All cause of mortality at 90-day and 12 months | 12 months
24-hours change in NIHSS (National Institutes of Health Stroke Scale) from baseline defined as the difference between NIHSS score at 24 hours and NIHSS score at admission. | 24 hours
  NIHSS (National Institutes of Health Stroke Scale) score is evaluated between 0-42 0 is normal and 42 maximal gravity
Subgroups analysis : Age (≤70 vs. >70 years) | 24 hours
Subgroups analysis :Baseline NIHSS≥10 vs NIHSS<10 (18) | 24 hours
Subgroups analysis : Volume of infarct area assessed by pc-ASPECTS (≤7 vs. >7) | 24 hours
  A pc-ASPECTS score of 10 indicates absence of visible ischemic changes in the posterior circulation, and pc-ASPECTS score of 0 indicates ischemic changes in the midbrain, pons, and bilateral thalami, posterior circulation territories, and cerebellar hemispheres
Subgroups analysis : Time from admission of patient in hospital to randomization (≤ 300 vs. > 300 minutes) | 360 minutes
Subgroups analysis: Baseline site of thrombi on vascular imaging (Top of the basilar artery vs other adjudicated by the core lab) | 24 hours
Subgroups analysis: Prior use of IV alteplase (yes vs. no) | 24 hours
Subgroups analysis : Collateral status (good versus poor, as adjudicated by the core lab on initial angiogram) with a 0-3 scale | 24 hours
  Collateral circulation is estimated by angiography with a 0-3 scale. The collateral status will be categorized as poor collaterals (scores 0-1) and good collaterals (scores 2-3)
Incidence of any intracerebral hemorrhage (ICH), parenchymal hematoma (PH), symptomatic ICH on brain imaging (Magnetic resonance imaging MRI or CT (computed tomography) scan) at 24±12h after thrombectomy (according to ECASS3 classification) | 24 hours
  ECASS III (European Cooperative Acute Stroke Study) classification :
  * Hemorrhage infarction type 1 (HI1)
  * Hemorrhage infarction type 2 (HI2)
  * Parenchymal hematoma type 1 (PH1)
  * Parenchymal hematoma type 2 (PH2)
Incidence of procedure-related complications defined as arterial perforation, arterial dissection, embolization in a new territory (ENT) and subarachnoid haemorrhage | hours
Cost-effectiveness analysis at 12 months | 12 months
  Incremental cost-effectiveness ratio (ICER, cost per quality-adjusted life year [QALY]), of Contact Aspiration (CA) first-line thrombectomy compared to standard first-line SR thrombectomy in treatment of AIS due to BAO, from a collective perspective and with a 12-months' time horizon.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo CONSOLI, Principal Investigator — Study principal investigator; Benjamin GORY, Study Chair — Scientific director
Locations (12):
- France (12):
  - Chu Bordeaux, Bordeaux
  - CHU Caen, Caen
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - Chru Nancy, Nancy
  - Chu Nantes, Nantes
  - APHP - Pitié Salpêtrière, Paris
  - Fondation Adolphe de Rothschild, Paris
  - CHU de Reims, Reims
  - CHU Rennes, Rennes
  - Hôpital FOCH, Suresnes
  - CHU de Tours, Tours